CLINICAL TRIAL: NCT07304219
Title: Physical Activity Based Treatment for Youth With Depression and Anxiety - a Pragmatic Randomized Controlled Trial
Brief Title: Physical Activity Based Treatment for Youth With Depression and Anxiety
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Western Norway University of Applied Sciences (Other); University of Bergen (Other); NORCE Norwegian Research Centre AS (Other)
Responsible Party: Principal Investigator, Arne Kodal, Researcher, NORCE Norwegian Research Centre AS
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 30912r
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Anxiety Depression
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: We will test the effectiveness of the CAHY intervention in a two-arm pragmatic randomized waitlist controlled trial (RCT) in which the participants will be randomly assigned to the intervention or the waitlist control group, following confirmation of eligibility and using a random number generator.
  Participants in the waitlist control group will be assigned to the intervention after the assessment at post-waitlist has been completed. The waitlist condition is of equal time-length as the intervention.
Who Masked: Participant, Care Provider
Masking Description: Randomization of participants is done by a random-number generator, and a mercantile ressource will allocate participants accordingly. Participants are not informed of the outcome of this randomization, and therapists providing the treatment are uanware of the randomization outcome.
  The primary investigator and outcomes assessor will know the result of the randomization, but have noe influence on the outcome of the randomization itself or allocation of participants to either condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): The Confident, Active and Happy-Youth intervention (CAHY), which is a group-based, bi-weekly, seven-week long, therapist-led intervention targeting core symptoms of anxiety and depression. Sessions are 50 mins. long, and offer a supportive, non-competitive, playful, and mastery-oriented climate to facilitate the individuals' need for relatedness, foster self-efficacy, motivation, fun and provide a safe space to practice exposure and gain positive experiences with social participation.Children and adolescents participate in age adjusted groups of max. eight: a child group age 8-10 years, a youngster group aged 11-3 years and adolescents group aged 14-17 years.
  Interventions: Behavioral: Confident, Active and Happy youth (CAHY)
- Waitlist Control (No Intervention): Participants randomized to this condition does not receive the intervention during the waitlist period, but receives CAHY intervention after the intervention i completed in the intervention group. Similar to the treatment group, they are measured before and after the waitlist period.

INTERVENTIONS:
Behavioral: Confident, Active and Happy youth (CAHY) — CAHY is a group-based, bi-weekly, seven-week long, therapist led intervention targeting core symptoms of anxiety and depression (barriers). Children and adolescents participate in age adjusted groups of max. eight: a child group age 8-10 years, a youngster group aged 11-3 years and adolescents group aged 14-17 years. Sessions are 50 mins. long, and offer a supportive, non-competitive, playful, and mastery-oriented climate to facilitate the individuals' need for relatedness, foster self-efficacy, motivation, fun and provide a safe space to practice exposure and gain positive experiences with social participation.
  CAHY incorporates established knowledge from physiological and psychological theory to address these barriers. The interventions targets youth with mental health disorders, and is delivered in a clinical setting.
  Arms: Treatment arm

SUMMARY:
The Confident, Active, and Happy Youth (CAHY) project aims to address the significant functional impairments experienced by youths with symptoms of depression and anxiety, focusing on physical activity (PA) and social participation. Traditional treatments, such as psychotherapy and pharmacotherapy, have shown moderate success, with many patients continuing to face functional and social challenges. This research seeks to fill that gap by testing the effectiveness of a physical activity-based intervention in a clinical setting to improve mental health and functional outcomes in clinical populations.

The study will be conducted as a pragmatic, randomized controlled trial, comparing CAHY with a waitlist control group in a real-world clinical setting. The intervention targets disease-specific barriers to PA and social participation, including fatigue, avoidance behaviors and low self-efficacy. The central challenge lies in adapting PA interventions to the clinical needs of youth with psychiatric disorders, which is essential for addressing the social and functional impairments associated with these disorders.

If proven effective, the results could have broad applications, offering a non-pharmacological treatment that is scalable and adaptable to various healthcare settings. The intervention supplements current treatment approaches and can improve patient outcomes in the short- and long-term, and can ultimately decrease healthcare service utilization by promoting better self-care and health habits

DETAILED DESCRIPTION:
The present research will examine the effectiveness of a novel supplemental intervention targeting children and adolescents with depression and anxiety symptoms. If proven efficacious, the research has broad applications in mental options; namely lack of physical activity, and interventions targeting functional outcomes in the form of social participation. and somatic healthcare.

Children and adolescents with depression and anxiety symptoms are significantly less physically active than their non-affected peers. Not only is PA vital to healthy development in children and adolescents, but low levels of physical activity are also significant risk factors for depression and anxiety, maintain, and aggravate these symptoms in children and adolescents. Physical activity is proven to be a low-cost, highly acceptable, non-stigmatizing intervention with no negative side-effects. Strong evidence indicates that physical activity is beneficial to mental health in youth in general and can be used in clinical populations towards mental health disorders such as depression and anxiety with moderate effect sizes. Towards long-term health trajectories, PA is a significant protective factor towards depression and anxiety specifically, mental and somatic diseases in general, and PA is also strongly related to overall lifespan. This translates to less service utilization (i.e. hospital and community services). Notably, PA is a modifiable factor in children and adolescents. However, PA is per today not included in treatment recommendations for youth mental health treatment (e.g. NICE guidelines) nor systematically used in child and adolescent treatment services.

Parallel to established knowledge of the health effects of adequate PA, social participation plays a crucial role in psychosocial development in children and adolescents. It fosters communication, empathy, teamwork, and conflict resolution, which are all vital skills in social settings and relationships including family, friendships, education, and work. Adolescents who are more socially engaged tend to have better long-term health trajectories (somatic and mental health), including higher levels of self-esteem, better social skills and well-being. Social participation is a primary factor in child and adolescents' functional level and youth with heightened depression and anxiety symptoms experience significant impairment in this area. Impairments in social participation are strongly linked to school absenteeism and dropout, loneliness, the development of chronic health conditions, and social exclusion. These outcomes represent a substantial societal challenge, one that the Norwegian government is actively working to address. Importantly, social participation is a modifiable factor and interventions specifically targeting this functional aspect of youths' mental health are limited.

Physical activity is commonly done in groups (i.e. football), and organized and non-organized physical activity (school or extracurricular) is a vital arena in terms of social training, social efficacy and social participation for children and adolescents. Thus, physical activity in groups provides a perfect platform and means to target depression and anxiety and address the social and functional impairments of depression and anxiety. Crucially, to unlock and make use of a physical activity based intervention in the treatment of youth depression and anxiety, it is paramount to address these youths disease- related barriers that deter them from using and joining in available physical and social opportunities, in their daily milieu. These barriers map onto the core symptoms of anxiety and depression; fatigue; low levels of physical activity; low confidence in one's ability to cope with situations that incite distress and/or fear; avoidance of engaging in situations that may incite distress and/or fear and lowered mood. For any intervention to be successful, it must specifically address and accommodate these barriers.

A major caveat with current research on physical activity and social participation falls on these barriers, which differentiates youth populations. Thus, findings from non-clinical populations with-out these barriers cannot be automatically taken to apply for clinical populations with these barriers. These is a paucity of studies examining the use of PA based interventions in clinical populations. Further, while a recent scoping-review of PA interventions in youth treated in child and adolescent mental health services (CAMHS) found evidence in support of the efficaciousness of PA towards depression and social participation, the review also indicated several limitations. Thus, numerous confounders were not controlled for including concurrent medication, co-morbid disorders, PA activity levels outside the intervention itself, and PA adherence in the intervention. Sample-sizes among included studies were low, many studies did not include control groups, and very few studies included assessment of psycho-social functioning. These limitations severely curb the conclusions that may be drawn and there is a lack of rigorous research on the topic.

The Confident, Active and Happy Youth Intervention Department of Child and Adolescent Mental Health Services (CAMHS), Haukeland University Hospital has in collaboration with users, developed and piloted a PA-based supplemental treatment, termed Confident, Active and Happy Youth (CAHY). The intervention targets children and adolescents with mental health disorders receiving treatment in CAMHS. The intervention targets core characteristics of depression and anxiety which constitute the barriers towards engaging in PA and social participation in the affected youth. The intervention addresses and accommodates the patients' -often ambivalent- motivation, lowered mood, high levels of avoidance and low levels confidence to engage in activities they seek to avoid.

2. Objectives and Goals/Milestones of the Project

Objectives and/or hypotheses It is the goal of this study, to establish the effectiveness of the Confident, Active and Happy Youth intervention, as a supplemental treatment for youth with mental health disorders, depressive and anxiety symptoms receiving treatment in Child and Adolescent Mental Health Care (CAMHS).

The study will be conducted as a pragmatic randomized controlled study, comparing active treatment to waitlist control. The study is pragmatic in that it is conducted in a real-world setting. Our research project aims to answer the following research questions:

* To what extent is the 7-week CAHY intervention successful in instigating the expected decrease in depressive and anxiety symptoms.
* What is the effectiveness of the CAHY-intervention towards instigating increased physical activity, increased social participation and quality of life in participants?
* What is the effectiveness of a physical activity intervention as a supplement to regular treatment in youths in treatment in CAMHS?
* What are the moderators of outcome for participants following a physical activity intervention?

The investigators hypothesize effects on the following primary outcomes compared to waitlist controls:

• Greater reduction in depressive and anxiety symptoms among participants.

The investigators hypothesize effects on the following secondary outcomes compared to waitlist controls:

* Improved quality of life and social participation.
* Improved daily PA.
* Improved social participation in community

The investigators expect intervention effects to be moderated by the following variables:

* Time spent in moderate-vigorous activity during and after the intervention.
* Severity of anxiety and depressive symptoms.
* Type and number of comorbid disorders.
* On-going treatment in CAMHS, (i.e. medication and/or psychotherapy).

Short and long-term goals A. Perform the RCT, B. Analyse data, C. Publish results, D. Disseminate results via research network and regional collaboration to relevant groups and new patient populations, E. Build a strong research group on the topic and develop PhD project(s) based on the study.

3. Methods 3.1. Study Design, Choice of Methodology and Analysis

The investigators will test the effectiveness of the CAHY intervention in a two-arm pragmatic randomized waitlist controlled trial (RCT) in which the participants will be randomly assigned to the intervention or the waitlist control group, following confirmation of eligibility and using a random number generator. Importantly, participants in the intervention and waitlist group have access to standard CAMHS care throughout the RCT, on the basis that this is their primary source of mental health care. It is not deemed ethical to withhold standard treatment for participants. Given that both intervention and waitlist groups continue with standard care, this will hinder any selection bias. Participants in the waitlist control group will be assigned to the intervention after the assessment at the post-intervention has been completed.

Study population and consent The target group are children and adolescents who receive healthcare treatment at a Child and adolescent specialized mental care clinic (CAMHS). Children and adolescents aged 8-17 are eligible.

Children and adolescents who should not do physical activity for health reasons are excluded.

Children and adolescents who do not wish or can not function in a group with other children and adolescents are excluded.

All participants in the study will be required to provide written consent. Informed written consent is obtained from all parents and assent is obtained from participants above age 12 years. Patients and parents can withdraw their consent at any time with no consequences for treatment in CAHY or CAMHS.

Measurements and outcomes

Primary outcomes:

- Anxiety symptoms and depression symptoms. The Revised Children's Anxiety and Depression Scale-25 (RCADS-25) is a 25-item scale that measures levels of anxiety (e.g. "I worry when I think I have done poorly at something") and low mood (e.g. "I feel sad or empty"). The scale has two subscales (Total Anxiety and Total Depression) and an overall score.

Secondary outcomes:

* Youth well-being. KID-SCREEN 27 is a generic questionnaire measuring health related quality of life and functional level.
* Social participation in community (school and extracurricular), child-, parent versions. Study pecific questionnaire assessing social participation in and outside school attendance.
* Daily physical activity level + session activity level: physical and sedentary activity (short and three-month follow-up). Objective measurement of activity using wearable activity sensor Actigraph GT3X+ monitor.
* Daily physical activity and sleep habits, parent interview. The Simple Physical Activity Questionnaire (SIMPAQ).

Other variables:

* Demographic data: Assessed with parent self-response questionnaire.
* Clinical characteristics: Participants give consent to access their CAMHS medical records.The investigators will retrieve following variables: a. CAMHS disorders, b. present medication, c. total time in CAMHS treatment before referral to CAHY, d. current CAMHS treatment offered (categorized).

Procedure Apart from participant's clinical characteristics, which will be manually collected from patient medical records following a codebook, assessments will be done digitally on a secure, research-approved platform, provided by Haukeland University Hospital. Participants are referred to the treatment by their attending therapist at one of the seven attending local outpatient Child and Adolescent Mental Health Clinic (CAMHS), Haukeland University Hospital. Referred and eligible participants are invited to a recruitment meeting where they receive detailed information about CAHY and the study and give consent/ascent to participate. Consenting participants fill out questionnaires at this time (T0). Enrolled participants are randomized to waitlist or active treatment and both receive login information to the study's digital platform. Prior to waitlist/treatment start, pre-assessment (T1) is made available on the platform, and post- and follow-up assessments are made available following treatment/waitlist end, and at 3 months post-treatment. Participants also are invited to a pre-treatment start-up consultation to familiarize themselves with the site and personnel, and a post-treatment consultation to summarize treatment learning points. Actigraphs will be provided to the participants in these pre- and post-treatment consultations. Participants will have their own actigraph, used in every session and throughout the study.

The Confident, Happy and Active Youth Intervention CAHY is a group-based, bi-weekly, seven-week long, therapist led intervention targeting core symptoms of anxiety and depression (barriers). Children and adolescents participate in age adjusted groups of max. eight: a child group age 8-10 years, a youngster group aged 11-3 years and adolescents group aged 14-17 years. Sessions are 50 mins. long, and offer a supportive, non-competitive, playful, and mastery-oriented climate to facilitate the individuals' need for relatedness, foster self-efficacy, motivation, fun and provide a safe space to practice exposure and gain positive experiences with social participation.

CAHY incorporates established knowledge from physiological and psychological theory to address these barriers and relies on three key components. Treatment effects of physical activity are obtained when participants engage in moderate to vigorous physical activity, defined by the energy expenditure of the task. The mechanisms span several neuro-biological and behavioral mechanisms and contribute to boost mood and reduce fatigue. The physical activity exposes the participants to behavioral activation and situations that are normally avoided. Participants are encouraged to engage with the feared stimuli fostering habituation (e.g., racing heart, social interaction, sweating etc.), learning and practicing new affective and cognitive regulation strategies (as opposed to avoidance). The physical activities provide participants with opportunities for autonomy and competence in interaction with others, thus addressing basic psychological needs, fostering self-efficacy and independence.

Personnel, equipment and setting The CAHY intervention is an available and fully funded treatment option for children and adolescents in Child and Adolescent Mental Health, Haukeland University Hospital. Four CAHY therapists are employed in CAMHs and have dedicated position earmarked CAHY. The therapists have different educational backgrounds: physiotherapy, psychiatric nurse, and a higher education in public health. Therapists will throughout the study be provided bi-weekly supervision by the study PI (Arne Kodal). The study is reliant on a part-time research assistant, whom will be funded by CAMHS. Digital infrastructure in the study is provided by Haukeland University Hospital and will be funded by the study. Actigraph instruments are lent from our collaborating research group, Physical Activity and Public Health, Western Norwegian University of Applied. Treatments sessions are delivered in the The Vitality Center for Children and Adolescents: (https://helse-bergen.no/avdelinger/energisenteret-for-barn-og-unge).

Power analysis

The following assumptions were applied in the calculation of sample size:

A moderate to large treatment effect, corresponding to Cohen's d between 0.50 and 0.80, is assumed to be detectable. Previous studies on the effects of group-based treatment for clinical samples of children and adolescents with anxiety and depressive symptoms have reported moderate to large effect sizes. TAG is a supplementary intervention to standard psychological and pharmacological treatment within Child and Adolescent Mental Health Services (CAMHS). Based on this, one could expect a supplementary treatment effect, where even a smaller effect size would be of clinical interest.

The intervention is delivered in groups of eight participants, which introduces a clustering effect that must be accounted for in the sample size calculation. A design adjustment for intra-class correlation (ICC) was therefore applied, with ICC set to 0.05, based on previous research on group-based interventions in mental health services. The correlation between measurement points (T1-T2) is estimated at r = 0.50, which increases the precision of the estimated change.

The sample size calculation was conducted in three steps:

1. Adjustment of the effect size for the correlation between measurement points according to the ANCOVA model.
2. Calculation of the required sample size per group using a two-sided t-test with significance level α = 0.05 and statistical power 1-β = 0.80.
3. Adjustment for the clustering effect using the design-effect formula:

DE=1+(m-1)⋅ICCDE = 1 + (m - 1)\cdot ICCDE=1+(m-1)⋅ICC where m is the number of participants per treatment group (here: 8).

Based on these assumptions, the required sample size for each of the two study arms (Intervention and Waitlist Control) is approximately 90 participants for a moderate effect size (Cohen's d = 0.50) and approximately 35 participants for a large effect size (Cohen's d = 0.80). This should be considered in light of recruitment capacity.

Data will be analyzed using SPSS version 26 and statistics program Stata and Mplus. Analyses of objective data on activity will be analyzed using Actilife software.

3.2 Organization and Collaboration The present research project is a collaboration between RKBU-Vest, Norce Research and Haukeland University Hospital. The CAHY-study was conceptualized by the main applicant, CAHY project leader, PhD and specialist in psychology Arne Kodal (arko@norceresearch.no/arne.kodal@helse-bergen.no), who is employed at both institutions. Kodal has led the feasibility trial of the intervention and together with the research group, outlined the proposed RCT. Kodal has broad clinical experience since 2006, holds a PhD in clinical psychology and did his thesis on a large RCT examining anxiety treatment in youths. Kodal's main research focuses on anxiety treatment and integration of physical activity in CAMHS. Kodal will be principal investigator in the study and responsible for the execution of the trial, first- or last-author main articles, develop PhD project(s) and lead all Work Packages (WP) 1-5.

CAHY Research Group consists of Professor Irene Elgen, Haukeland University Hospital: specialist in child pediatrics and psychiatry with extensive knowledge on the interplay between mental and somatic health, Professor Kjell Morten Stormark, Norce Research: expert on child and adolescent development, epidemiological research and research designs, Professor Gro Janne Wergeland, University of Bergen: expert on anxiety treatment and clinical-trial assessment, Professor Eivind Aadland, Western Norway University of Applied Sciences: expert on objective measurement of PA in children, adolescents and adults. Assistant Professor Lars Peder Vatshelle Bovim, is leader of the Childrens Vitality Center and PI on the sister project to CAHY, "Mestringsuker".

Research-group collaboration. This project is a collaboration between a clinical unit at the Child and Adolescent Mental Health, Division of Psychiatry, Haukeland University Hospital (HUH), and three research groups. These groups are the Child and Adolescent Research Group at CAMHS, HUH, led by Professor Irene Elgen; Public Mental Health Research Group at the Regional Centre for Child and Youth Mental Health and Child Welfare, part of the Norwegian Research Centre (NORCE), headed by Professor Kjell Morten Stormark; Physical Activity and Public Health, Western Norwegian University of Applied Science led by Professor Eivind Aadland. As advocates for developing evidenced-based programs for youths in the mental health sector, research groups at CAMHS and Norce and the clinical unit at Haukeland have extensive expertise in implementing and executing RCTs to evaluate intervention effectiveness. Aadland and his research group, are leading Norwegian experts on the impact of PA on health and objective measurement of PA, heading numerous studies on the topic. Aadland and his group provide measurement equipment and methodology expertise to assess objective PA levels in our population.

Vitality Center research collaboration. The CAHY study is also firmly anchored in the Childrens Vitality Center, HUH, which spans mental-somatic healthcare. The center has spawned several associated projects, the closest of which is currently undergoing feasability testing ("Mestringsuker": https://www.helse-bergen.no/avdelinger/barne-og-ungdomsklinikken/energisenteret/mestringsuker/). The Vitality Center is also at the root of an initiative to establish a new research center for children's health, "Forskningssenter for Barnehelse", focusing on children's health in life-course perspective. The CAHY model of treatment, is integrated in and aligned with this initiative.

Project NGO collaboration is established with the Council for Mental Health and Senior Advisor, Werner Fredriksen. He is leader of the Norwegian National Network for Exercise in Treatment. Fredriksen will be a key player in the dissemination of results to national networks of healthcare professional.

3.4. Plan for Milestones and Dissemination

Main planned study publications are:

* Physical activity and social participation: diagnostic characteristics of children and adolescents in mental health care outpatient clinics. The article examines diagnostic, physical activity, inactivity, social participation and functional characteristics of youth treated in CAMHS.
* Effectiveness of a physical activity intervention for children and adolescents with anxiety and depression, treated in CAMHS - a randomized controlled trial. The article reports on the main findings of our study in terms of treatment outcomes.
* Moderators of outcomes of a physical activity intervention for children and adolescents with anxiety and depression, treated in CAMHS. The article examines moderators of treatment outcome.
* Development of a moderate to vigorous physical activity intervention for youths in treatment for mental health disorders: a co-creation prosses between users, clinicians and researchers. The article details the co-creative process of the development, and implementation of CAHY in mental health care.

Additional publications are planned and will examine trajectories of psychological needs, well-being, self-efficacy changes and their influence on social and PA participation. The investigators seek to develop these research questions into a separate PhD project, within the CAHY project, thus strengthening our research group.

CAHY results will be disseminated in leading international peer reviewed journals. The investigators will disseminate results together with our collaborating research groups, users and the Council for Mental Health (Rådet for Psykisk Helse) targeting broader audiences through various outlets, international and national conferences, chronicles, newspapers articles and public lectures.

3.5 Plans for Implementation The CAHY intervention is already implemented as an available treatment option for children and adolescents in Child and Adolescent Mental Health, Haukeland University Hospital, although a thorough assessment of effectiveness is lacking - hence the aim of this study. If proven successful, the intervention will continue as an available treatment option for youths in CAMHS, but the investigators will also build on results and further develop the approach and research, i.e. new patient groups, intensive version, investigation of specific mechanisms. The study will also provide valuable corroborative data to our sister project, Mestringsuker, thus providing support for broader exploitation of a PA based intervention in general specialized healthcare. Our collaboration with the Childrens Vitality Center will promote further exploitation of results in broader pediatric populations, including somatic healthcare, many of whom share the same impairments and barriers to PA and social participation.

3.6 Risk Management Our feasibility trial revealed no adverse effects of the intervention, and other studies using physical activity interventions have found no negative side-effects of such interventions. Importantly, as this is an add-on treatment, the participants continue to have access to ongoing treatment in CAMHS, either they complete or drop-out of the CAHY intervention. In terms of participant recruitment issues, our feasability study revealed no such challenges. Additionally, continuous monitoring of intervention capacity and incoming referrals is in place, and referrals can be increased via information channels within the clinic, including available websites, meetings between CAHY staff and clinics, flyers and poster in all participating clinics.

The intervention itself is funded and delivered in the premises of the Childrens Vitality Center, by CAHY therapists. The infrastructure and necessary equipment to implement the RCT is in place. The feasibility study indicated the need for slight changes to treatment protocol. These changes to protocol have been undertaken in 2024-25, and relevant changes have been approved by the Regional Ethics board.

5. Ethical Considerations The Regional Committee for Medical Research Ethics has approved the study (ID Number: 30912) and study end-date is set for mid 2028. The study will be performed in accordance with the national and local regulatory requirements. The study will be registered in clnicaltrials.org. None of the assessments involve any health risk, and the investigators believe most participants will benefit from participation in the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to treatment for psychiatric disorder at the Child and Adolescent Mental Health Services at Haukeland University Hospital (Psykisk helsevern for barn og unge, Helse Bergen)

Exclusion Criteria:

* The CAHY treatment is contraindicated (e.g. in severe eating disorders)
* When participation would compromise the benefit for other patients in the group

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
The Revised Child Anxiety and Depression Scale (RCADS) | From enrollment to follow-up three months after end of treatment
  The Revised Children's Anxiety and Depression Scale-25 (RCADS-25) is a 25-item scale that measures levels of anxiety (e.g. "I worry when I think I have done poorly at something") and low mood (e.g. "I feel sad or empty"). The scale has two subscales (Total Anxiety and Total Depression) and an overall score.

SECONDARY OUTCOMES:
Kidscreen-27 | From enrollment to follow-up three months after end of treatment
  The KID-SCREEN 27 (Ravens-Sieberer et al., 2007) is a generic questionnaire measuring health related quality of life and functional level.
Participation in community | From enrollment to follow-up three months after end of treatment
  This is a project-specific instrument, aimed at measuring youths social participation in community arenas such as school, extracariccular activities, engagement in physical activity and social relations. The questionnaire is a 17 question long, multiple choice questionnaire.
Objective physical activity | From enrollment to follow-up three months after end of treatment
  Participants physical activity, will be objectively measured by means of an electronic, wearable activity monitor.
Simple Physical Activity Questionnaire | From enrollment to follow-up three months after end of treatment
  The Simple Physical Activity Questionnaire (SIMPAQ) (Rosenbaum et al., 2020) is a short,, structured, interview based questionnaire, assessing participants daily physical activity and sleep habits.

CONTACTS AND LOCATIONS:
Overall Officials: Arne Kodal, PhD, Principal Investigator — NORCE - Norwegian Research Centre
Locations (1):
- Haukeland University Hospital, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: Undecided